CLINICAL TRIAL: NCT01979640
Title: Adequate Additional Bronchial Cuff Volume to Achieve Blood-tight Seal After Air-tight Seal in Double Lumen Tube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHBahk_DLT_bloodtightseal
Record Dates: First submitted 2013-11-03; First posted 2013-11-08 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Preventing Blood Leakage of Bronchial Cuff
Keywords: bronchial cuff; double lumen tube; blood tight seal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 39 Fr double lumen group (Experimental): patients are assigned to 35 Fr, 37 Fr, 39 Fr double lumen tube group according to their left main bronchus diameter measured by preoperative chest CT, to minimize difference between main bronchus diameter and bronchial tip diameter of double lumen tube
  Interventions: Procedure: 39 Fr double lumen tube group
- 37 Fr double lumen group (Experimental): patients are assigned to 35 Fr, 37 Fr, 39 Fr double lumen tube group according to their left main bronchus diameter measured by preoperative chest CT, to minimize difference between main bronchus diameter and bronchial tip diameter of double lumen tube
  Interventions: Procedure: 37 Fr double lumen tube group
- 35 Fr double lumen tube group (Experimental): patients are assigned to 35 Fr, 37 Fr, 39 Fr double lumen tube group according to their left main bronchus diameter measured by preoperative chest CT, to minimize difference between main bronchus diameter and bronchial tip diameter of double lumen tube
  Interventions: Procedure: 35 Fr double lumen tube group

INTERVENTIONS:
Procedure: 39 Fr double lumen tube group — additional bronchial cuff volume is decided according to up-and-down biased coin design sequential method, by incremental volume of 0.1 ml
  Arms: 39 Fr double lumen group
Procedure: 37 Fr double lumen tube group — additional bronchial cuff volume is decided according to up-and-down biased coin design sequential method, by incremental volume of 0.1 ml
  Arms: 37 Fr double lumen group
Procedure: 35 Fr double lumen tube group — additional bronchial cuff volume is decided according to up-and-down biased coin design sequential method, by incremental volume of 0.1 ml
  Arms: 35 Fr double lumen tube group

SUMMARY:
The purpose of this study is to find the adequate additional bronchial cuff volume after achievement of air-tight seal, that can achieve blood-tight seal(preventing leakage of blood through cuff) in double lumen tube

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thoracic surgery under left lower decubitus position, using left sided double lumen tube
* patient's left main bronchus size adequate for 35Fr, 37 Fr, 39 Fr double lumen tube

Exclusion Criteria:

* dislocation or great movement of double lumen tube depth

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
leakage of autologus blood through bronchial cuff | 10, 20, 30 minutes after dripping of blood around bronchial cuff

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea